CLINICAL TRIAL: NCT01224002
Title: A Comparative Feasibility Study to Assess the Prevalence and Severity of Dental Caries in Incarcerated People Who Abuse Methamphetamine
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910215; 10-D-N215
Record Dates: First submitted 2010-10-16; First posted 2010-10-19 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Substance-Related Disorders; Dental Caries
Keywords: Cross-Sectional; Observational; Comparative; Retrospective; Feasibility; Dental Decay; Drug Abuse; Survey
MeSH Terms: conditions — Substance-Related Disorders; Dental Caries

SUMMARY:
The prevalence and severity of dental caries in incarcerated people who abuse drugs are unknown but an inmate reporting to the dental clinic typically presents with myriad findings: oral signs of uncontrolled decay on the buccal smooth surfaces of the posterior teeth and interproximal surfaces of the anterior teeth, excessive tooth wear due to grinding and clenching, and gingival inflammation. The primary risk factors for the development of caries appear to be the combination of xerostomia, frequent consumption of carbonated soft drinks, high dental plaque levels and nonexistent or inadequate oral hygiene. Since some of these findings are seen in the other disease states, specifically in substance abuse cases, the diagnosis is often not clear. The objective of the project is to design a cross sectional comparative feasibility study that will estimate the prevalence, pattern, and severity of untreated dental decay for three types of inmates: methamphetamine abusers, substance abusers not identified as methamphetamine users, and non-substance abusers, focusing in on methamphetamine abusers as the highest risk group.

Recruitment will be accomplished using a 2-phased process. Phase I. An invitation letter explaining the study purpose and its relevance to oral health in a correctional setting will be mailed to the inmate population at two Federal Bureau of Prisons' institutions who entered the prison system during the first half of 2009. Dublin, a female FCI located in Northern California and Butner, a male FCC located in North Carolina were the selected facilities due to the high incidence of drug abusers among their inmates. The letter, which will invite all inmates to participate in the study, will inform the inmate should they consent to participate in the study that they will have their existing dental record confirmed, Central File reviewed for DSM-IV diagnosis pertinent to the study, and that they will be given a study questionnaire. Positive responses to the invitation letters will be returned to Dr. Johnson at head quarters in Washington DC. The psychology division will code the volunteer inmates into the three study groups.

Phase II. The first 30 chronologically documented volunteers in each study group category will be scheduled an appointment. A consent form will be read and explained to each inmate, in either English or Spanish as appropriate and his/her signature obtained as his/her informed consent.

Each question on the study questionnaire will be read to the inmate volunteer and the Research Associate will record the answer. A retrospective comparative study will then be employed utilizing the inmate's initial dental intake exam (routinely administered by the Federal Bureau of Prisons' dental department). The dental chart will be abstracted for dental caries. The pattern of surface-specific dental caries (DFS index) will be described and analyzed. The focus will be on the levels of untreated and treated disease diagnosed in a 4-zone partition of the oral dentition, representing a modification of the zones identified in the Grainger's caries severity index scoring system as this partition allows focus on decay patterns of anterior tooth surfaces. The multivariate summary of disease levels within each zone will be derived and statistically compared across the three study groups using Hotelling's t2-test (the multivariate extension of the Student-t test). The results of the study will be used to do a preliminary assessment between methamphetamine drug abuse and oral health and determine whether a prospective clinical study is warranted.

DETAILED DESCRIPTION:
The prevalence and severity of dental caries in incarcerated people who abuse drugs are unknown but an inmate reporting to the dental clinic typically presents with myriad findings: oral signs of uncontrolled decay on the buccal smooth surfaces of the posterior teeth and interproximal surfaces of the anterior teeth, excessive tooth wear due to grinding and clenching, and gingival inflammation. The primary risk factors for the development of caries appear to be the combination of xerostomia, frequent consumption of carbonated soft drinks, high dental plaque levels and nonexistent or inadequate oral hygiene. Since some of these findings are seen in the other disease states, specifically in substance abuse cases, the diagnosis is often not clear. The objective of the project is to design a cross sectional comparative feasibility study that will estimate the prevalence, pattern, and severity of untreated dental decay for three types of inmates: methamphetamine abusers, substance abusers not identified as methamphetamine users, and non-substance abusers, focusing in on methamphetamine abusers as the highest risk group.

Recruitment will be accomplished using a 2-phased process. Phase I. An invitation letter explaining the study purpose and its relevance to oral health in a correctional setting will be mailed to the inmate population at two Federal Bureau of Prisons' institutions who entered the prison system during the first half of 2009. Dublin, a female FCI located in Northern California and Butner, a male FCC located in North Carolina were the selected facilities due to the high incidence of drug abusers among their inmates. The letter, which will invite all inmates to participate in the study, will inform the inmate should they consent to participate in the study that they will have their existing dental record confirmed, Central File reviewed for DSM-IV diagnosis pertinent to the study, and that they will be given a study questionnaire. Positive responses to the invitation letters will be returned to Dr. Johnson at head quarters in Washington DC. The psychology division will code the volunteer inmates into the three study groups.

Phase II. The first 30 chronologically documented volunteers in each study group category will be scheduled an appointment. A consent form will be read and explained to each inmate, in either English or Spanish as appropriate and his/her signature obtained as his/her informed consent.

Each question on the study questionnaire will be read to the inmate volunteer and the Research Associate will record the answer. A retrospective comparative study will then be employed utilizing the inmate's initial dental intake exam (routinely administered by the Federal Bureau of Prisons' dental department). The dental chart will be abstracted for dental caries. The pattern of surface-specific dental caries (DFS index) will be described and analyzed. The focus will be on the levels of untreated and treated disease diagnosed in a 4-zone partition of the oral dentition, representing a modification of the zones identified in the Grainger's caries severity index scoring system as this partition allows focus on decay patterns of anterior tooth surfaces. The multivariate summary of disease levels within each zone will be derived and statistically compared across the three study groups using Hotelling's t2-test (the multivariate extension of the Student-t test). The results of the study will be used to do a preliminary assessment between methamphetamine drug abuse and oral health and determine whether a prospective clinical study is warranted.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Inmates who have undergone medical, dental and psychological evaluation during their intake into the Butner or Dublin facilities between January 2010 and December 2010.
* Age between 18 and 65.
* At least 16 existing natural teeth, root tips included. The reason for choosing this relatively high number is in order to have sufficient data for an analysis of patterns of decay.

EXCLUSION CRITERIA:

* History of head and neck radiation therapy as documented by health history
* History of Sjogren's syndrome or similar exocrine disorders, as documented by health history
* Currently in active orthodontic treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Study Completion 2012-11

CONTACTS AND LOCATIONS:
Overall Officials: J. Silvio Gutkind, Ph.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)

REFERENCES:
- [Background] Shaner JW. Caries associated with methamphetamine abuse. J Mich Dent Assoc. 2002 Sep;84(9):42-7. PMID 12271905
- [Background] Klasser GD, Epstein J. Methamphetamine and its impact on dental care. J Can Dent Assoc. 2005 Nov;71(10):759-62. PMID 16324229
- [Background] Donaldson M, Goodchild JH. Oral health of the methamphetamine abuser. Am J Health Syst Pharm. 2006 Nov 1;63(21):2078-82. doi: 10.2146/ajhp060198. PMID 17057044